CLINICAL TRIAL: NCT02104115
Title: Effects of Bread Gluten Content on Gastrointestinal Volumes
Acronym: EGG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: E12122013 SoM NDDC EEG
Record Dates: First submitted 2014-03-25; First posted 2014-04-04 (Estimated); Last update posted 2015-10-06 (Estimated); Status verified 2015-10

CONDITIONS: Healthy
Keywords: Stomach; Small bowel; Colon; MRI; Function; Gastrointestinal volumes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Gluten free white bread (Other): Sliced loaf of gluten free white bread
  Interventions: Other: MRI scanners; Other: VAS Symptom scores
- Normal gluten content white wheat bread (Other): Sliced loaf of normal gluten content white wheat bread
  Interventions: Other: MRI scanners; Other: VAS Symptom scores
- High gluten content white wheat bread (Other): Sliced loaf of high gluten content white wheat bread
  Interventions: Other: MRI scanners; Other: VAS Symptom scores

INTERVENTIONS:
Other: MRI scanners
Other: VAS Symptom scores

SUMMARY:
The investigators will apply non invasive Magnetic Resonance Imaging (MRI) techniques developed in Nottingham to evaluate the gastric emptying, small bowel water content, colonic gas and volumes in healthy volunteers eating three breads with different amount of gluten (none, normal, or high gluten) in three consecutive weeks.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-55
* Able to give informed consent

Exclusion Criteria:

* Unable to abstain from smoking for the duration of the study
* Pregnancy declared by candidate
* History declared by the candidate of pre-existing gastrointestinal disorder, including but not limited to: Inflammatory Bowel Disease, Coeliac Disease, Pancreatitis, Gallstone disease (biliary colic, cholecystitis), Diverticulitis, Cancer of the gastrointestinal tract, Irritable Bowel Syndrome
* Reported history of previous resection of any part of the gastrointestinal tract other than appendix or gallbladder
* Any medical condition making participation potentially compromising participation in the study e.g. diabetes mellitus, respiratory disease limiting ability to lie in the scanner
* Contraindications for MRI scanning i.e. metallic implants, pacemakers, history of metallic foreign body in eye(s) and penetrating eye injury
* Reported alcohol dependence
* Taking any drug known to alter GI motility including mebeverine, opiates, monoamine oxidase inhibitors, phenothiazines, benzodiazepines, calcium channel antagonists during or in the 2 weeks prior to the test. (Selective serotonin reuptake inhibitors and low dose tricyclic antidepressants will be recorded but will not be an exclusion criteria)
* Antibiotic or probiotic treatment in the past 4 weeks
* Inability to lie flat or exceed scanner limits of weight <120kg
* Poor understanding of English language
* Participation in night shift work the week prior to the study day. Night work is defined as working between midnight and 0600
* Strenuous exercise greater than 10 hours per week (i.e. no competition training the week prior to the study).
* Participation in any medical trials for the past 3 months
* Anyone who in the opinion of the investigator is unlikely to be able to comply with the protocol e.g. cognitive dysfunction, chaotic lifestyle related to substance abuse

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2014-03; Primary Completion 2014-07 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Change in gastric volume from baseline to 360 minutes after feeding | baseline and 0, 60, 120, 180, 240, 300, 360 minutes after feeding

SECONDARY OUTCOMES:
Change in small bowel water content from baseline to 360 minutes after feeding | baseline and 0, 60, 120, 180, 240, 300, 360 minutes after feeding

OTHER OUTCOMES:
Change in colonic total volume from baseline to 360 minutes after feeding | baseline and 0, 60, 120, 180, 240, 300, 360 minutes after feeding
Change in VAS for symptom scores (fullness, hunger, desire to eat, bloating, nausea, abdominal discomfort / pain) from baseline to 360 minutes after feeding | baseline, 0, 60, 120, 180, 240, 300, 360 minutes after feeding
Change in colonic gas volumes from baseline to 360 minutes after feeding | baseline and 0, 60, 120, 180, 240, 300, 360 minutes after feeding

CONTACTS AND LOCATIONS:
Overall Officials: Marina Coletta, Fellow in Gastroenterology, Principal Investigator — Visiting fellow in Gastroenterology; Luca Marciani, Lecturer, Principal Investigator — Lecturer in Gastrointestinal Imaging; Robin Spiller, Professor, Study Director — Professor of Gastroenterology; Giles Major, Fellow, Principal Investigator — University of Nottingham; Gemma Chaddock, BSc, Principal Investigator — University of Nottingham
Locations (2):
- United Kingdom (2):
  - Sir Peter Mansfield Magnetic Resonance Centre, University of Nottingham, Nottingham
  - Nottingham Digestive Diseases Centre, E floor West Block, QMC Campus, Nottingham University Hospitals, Nottingham

REFERENCES:
- [Background] Marciani L. Assessment of gastrointestinal motor functions by MRI: a comprehensive review. Neurogastroenterol Motil. 2011 May;23(5):399-407. doi: 10.1111/j.1365-2982.2011.01670.x. Epub 2011 Jan 30. PMID 21276139
- [Background] Marciani L, Pritchard SE, Hellier-Woods C, Costigan C, Hoad CL, Gowland PA, Spiller RC. Delayed gastric emptying and reduced postprandial small bowel water content of equicaloric whole meal bread versus rice meals in healthy subjects: novel MRI insights. Eur J Clin Nutr. 2013 Jul;67(7):754-8. doi: 10.1038/ejcn.2013.78. Epub 2013 Apr 17. PMID 23594839
- [Background] Lobo DN, Hendry PO, Rodrigues G, Marciani L, Totman JJ, Wright JW, Preston T, Gowland P, Spiller RC, Fearon KC. Gastric emptying of three liquid oral preoperative metabolic preconditioning regimens measured by magnetic resonance imaging in healthy adult volunteers: a randomised double-blind, crossover study. Clin Nutr. 2009 Dec;28(6):636-41. doi: 10.1016/j.clnu.2009.05.002. Epub 2009 Jun 4. PMID 19500889
- [Background] Hoad CL, Marciani L, Foley S, Totman JJ, Wright J, Bush D, Cox EF, Campbell E, Spiller RC, Gowland PA. Non-invasive quantification of small bowel water content by MRI: a validation study. Phys Med Biol. 2007 Dec 7;52(23):6909-22. doi: 10.1088/0031-9155/52/23/009. Epub 2007 Nov 8. PMID 18029983
- [Background] Marciani L, Cox EF, Hoad CL, Pritchard S, Totman JJ, Foley S, Mistry A, Evans S, Gowland PA, Spiller RC. Postprandial changes in small bowel water content in healthy subjects and patients with irritable bowel syndrome. Gastroenterology. 2010 Feb;138(2):469-77, 477.e1. doi: 10.1053/j.gastro.2009.10.055. Epub 2009 Nov 10. PMID 19909743